CLINICAL TRIAL: NCT04802850
Title: Investigation of Immediate, Short and Long Term Effects of Mulligan Mobilization With Movement Techniques in Nonspesific Chronic Low Back Pain: a Randomized Placebo-controlled Trial
Brief Title: Investigation of Immediate, Short and Long Term Effects of Mulligan Mobilization With Movement Techniques in Nonspesific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, HATİCE YAKUT, principal investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: study1984
Record Dates: First submitted 2021-03-06; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Movement

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real MWM (Experimental): Real mobilization with movement
  Interventions: Other: Mulligan mobilization with movement
- Sham MWM (Sham Comparator): sham or placebo mobilization with movement
  Interventions: Other: Mulligan mobilization with movement

INTERVENTIONS:
Other: Mulligan mobilization with movement

SUMMARY:
Introduction: Although the effectiveness of many mobilization methods in chronic low back pain (CLBP) was shown, these effects were not monitored in the long term. The aim of this study was to identify the immediate, short and long-term effects of mulligan mobilization with movement (MWM) in terms of pain, range of motion (ROM), flexibility, endurance, functionality and disabilities in patients with CLBP. Methods: The study was designed in randomized-placebo controlled with 36 people randomly distributed into 2 groups. Sustained natural apophyseal glide (SNAG) was applied to the lumbar region, straight leg raise (SLR) with traction to the hip, and internal rotational mobilization techniques and home exercise program were applied in Group 1 (n=19); and the same techniques were applied as sham mobilization in Group 2 (n=17). The evaluations were made as post-intervention for immediate effect, and were also made at the 5th week, 3rd month, and 6th months for short and long-term effect. Evaluation was also made for pain in 12th month.

ELIGIBILITY:
Inclusion Criteria:

* Having 3 months' continuous or intermittent LBP symptoms, without leg pain above the knee
* Pain at VAS > 3/10,
* Back pain increased by active lumbar flexion movement

Exclusion Criteria:

* Confirmed nerve root compression
* Neurological symptoms
* Lumbar spine stenosis
* Back surgery history
* Chronic pain syndrome
* LBP from fracture
* Infection
* Visceral disease
* Pregnancy
* Major clinical depression
* Cauda equina syndrome
* Significant osteoporosis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Flexibility | immediate(post intervention)-5 weeeks(after 5 week treatment)-3 months(after 3 months)-6 months(after 6 months)
  Change of lumbar flexibility with sit and reach objective test( cm)
Endurance | immediate(post intervention)-5 weeeks(after 5 week treatment)-3 months(after 3 months)-6 months(after 6 months)
  Change of endurance of lumbar extensors with Sorensen endurance test(sn)
Functionality with patient specific function scale | immediate(post intervention)-5 weeeks(after 5 week treatment)-3 months(after 3 months)-6 months(after 6 months)
  Change of function
Disabilities with Oswestry disability index(scale) | immediate(post intervention)-5 weeeks(after 5 week treatment)-3 months(after 3 months)-6 months(after 6 months)
  Change of disabilities

SECONDARY OUTCOMES:
range of motion with goniometer | immediate(post intervention)-5 weeeks(after 5 week treatment)-3 months(after 3 months)-6 months(after 6 months)-12 months
  change of range of motion

IPD SHARING:
Plan to Share IPD: Undecided